CLINICAL TRIAL: NCT01771536
Title: The PCI Choice Trial: a Pilot Randomized Trial of a Decision Aid for Patients With Stable Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-004554
Record Dates: First submitted 2012-12-15; First posted 2013-01-18 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI Choice decision (Active Comparator): Decision Aid intervention is provided to clinician to share with patient
  Interventions: Other: Decision Aid
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Decision Aid
  Arms: PCI Choice decision

SUMMARY:
Despite several large clinical trials clearly establishing that coronary revascularization (i.e. percutaneous coronary intervention - PCI) does not prolong survival or prevent myocardial infarction (MI) for stable coronary artery disease (CAD), patients with stable angina continue to believe that PCI is performed to improve these outcomes. Additionally, recent concerns have emerged of overuse of PCI among patients with little or no angina. Thus there is a compelling need to share with patients the risks and benefits of PCI prior to treatment to reach an informed decision.

This study is designed to answer the question of whether a decision aid can improve patient knowledge, decisional conflict and patient satisfaction with decision-making compared to usual care for the treatment of stable angina.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stable angina - As judge by clinician, eligible for medication therapy or PCI - agree to be available for follow-up survey 3 months after treatment decision

Exclusion Criteria:

* has major communication barrier (severe hearing/vision impairment, dementia, cannot communicate with clinician in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of the PCI Choice Decision aid vs. Usual Care assessed by Patient and Provider Surveys, and encounter Video/Audio Recordings | Baseline to Three Months
  Efficacy in improving measures of patient knowledge and involvement, decision making quality, treatment choice and clinician satisfaction of the decision aid.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Shah, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Coylewright M, Dick S, Zmolek B, Askelin J, Hawkins E, Branda M, Inselman JW, Zeballos-Palacios C, Shah ND, Hess EP, LeBlanc A, Montori VM, Ting HH. PCI Choice Decision Aid for Stable Coronary Artery Disease: A Randomized Trial. Circ Cardiovasc Qual Outcomes. 2016 Nov;9(6):767-776. doi: 10.1161/CIRCOUTCOMES.116.002641. Epub 2016 Nov 1. PMID 27803090
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials